CLINICAL TRIAL: NCT00322478
Title: Non-Significant Risk Investigational Device Study of the Wireless GlucoMON™ Glucose Meter Accessory and Real-time Blood Glucose Alerts as an Enabling Technology for People Who Team Manage Diabetes
Brief Title: Diabetes Technology Study of Real-Time Glucose Alerts in the Team Management of Diabetes
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Diabetech (Industry)
Responsible Party: Principal Investigator, Kevin L. McMahon, Principal Investigator, Diabetech
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: DIRB1-2006-1
Record Dates: First submitted 2006-05-05; First posted 2006-05-08 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-10

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GlucoMON-ADMS enabled (Other): Patients who are equipped with the automated technology vs. standard/conventional care
  Interventions: Behavioral: Automated informatics driven education and social networking; Behavioral: Blood Glucose Notifications to Remote Caregivers; Behavioral: Frequency of Pattern Management

INTERVENTIONS:
Behavioral: Automated informatics driven education and social networking — The patient uses a self-contained wireless accessory to a standard blood glucose meter. This device manages the meter to ensure accurate time stamps and transmits the data to a centralized data management system. The system is then configured to assess the data and take automated steps to derive relevant diabetes education and/or send reports to a registered and authorized team.
  Other Names: The GlucoMON GSM/GPRS Appliance - NSR Investigational Device
Behavioral: Blood Glucose Notifications to Remote Caregivers — When children with type 1 diabetes are at school they will connect their blood glucose meter to the GlucoMON appliance. The data from the meter is then transmitted to the central system followed by the most recent blood sugar being sent to the primary caregiver's email address(es) as a plain text message. The investigator is interested to better understand the behaviors that accompany the expectation of the message and actions taken subsequent to receipt of the message by the patient-centric team.
  Other Names: School Day Diabetes Management
Behavioral: Frequency of Pattern Management — The behavioral intervention being studied involves the assessment of frequency of self-care in relation to the primary and secondary outcomes including overall blood sugar control and patient satisfaction.
  Other Names: Automated blood sugar pattern management; Day over Day blood sugar report

SUMMARY:
Many people with diabetes have a desire to share blood glucose data with other members of their team. Using a unique wireless glucose meter device, real-time wireless alerts may be automatically sent to a specific team of interested caregivers whom the patient selects. Additionally, trending reports can be automatically delivered to any number of authorized patient caregivers to facilitate more frequent review of glycemic control.

This study is recruiting patients from throughout the USA including Hawaii and Alaska.

DETAILED DESCRIPTION:
Previous research suggests that using wireless messaging to handle the values from finger-stick blood glucose testing and making the numbers available to both patients and their diabetes health care team may improve the management of diabetes. We would like to test the GlucoMON glucose meter accessory device and the real-time wireless alerts feature which automatically sends to a specific team of interested caregivers whom the patient selects and the effects of real-time alerts in the management of diabetes. We also would like to know whether this procedure can improve the frequency of glucose pattern management as a patient and possibly reduce the costs of care required for frequent interactions between the patient and the diabetes care team.

In this study, we will compare a new wireless device and Internet-based automated data management system to existing methods of sharing data amongst an interested care team. Specifically, the research will answer the question, "How does the real-time alert feature of the GlucoMON device compare to people who regularly initiate telephone calls (notification) to interested members of the care team to report a) that a blood glucose test was performed; b) the numerical value of the blood glucose level; and, c) the time that the blood glucose test was performed?" In addition, the data collected during this study will be used to answer the larger question of whether the automated sharing of patient directed blood sugar information affects diabetes control positively or negatively and to what degree.

The GlucoMON device provided by Diabetech, LP is an automated, wireless blood glucose collection and reporting system that will be used to send encrypted glucose data through a secure Internet connection for review by the patient and the authorized diabetes care team. Preparing and delivering the glucose data in this manner will help the care team to know if the person with diabetes is testing or not and provide them with some level of information regarding current blood glucose control even though they cannot be with the patient.

The most obvious use of this feature of the automated diabetes management system is the delivery of a blood sugar text message to the mother and/or father of a child with type 1 diabetes attempting to provide remote assistance to their son or daughter at school. However, this is only one scenario in which the researchers anticipate patient feedback.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent/Assent Form Completion including signature(s) required prior to final enrollment
* Previously diagnosed with diabetes (any type)
* Participant must be willing to subsidize a portion of the cost of the research by agreeing to a participant fee

Exclusion Criteria:

* Since the study device depends on nationwide wireless network coverage, only those patients who reside within the wireless network coverage area will be allowed to participate in this study. The Investigator will confirm adequate coverage based on zip code prior to enrollment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2006-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Blood Sugar Control | Daily and Quarterly
Patient Satisfaction | Quarterly

SECONDARY OUTCOMES:
A1c | Quarterly
Self-Test Frequency of SMBG | Daily
Standard Deviation of A1c and SMBG | Daily via MAGE if eligible for analysis

CONTACTS AND LOCATIONS:
Overall Officials: Kevin L McMahon, BS, Principal Investigator — Sponsor-Investigator
Locations (1):
- Diabetech, Dallas, Texas, United States